CLINICAL TRIAL: NCT07398339
Title: A Multicenter, Open-Label, Phase IIa Clinical Study Evaluating the Preliminary Efficacy and Safety of Sodium Porphyrin Injection Combined With Photodynamic Therapy Plus Gemcitabine and Cisplatin Chemotherapy in Patients With Advanced Extrahepatic Cholangiocarcinoma With Biliary Obstruction
Brief Title: Cosiporfin Sodium for Injection Photodynamic Therapy
Acronym: DVDMS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Guangsheng Biopharmaceutical Co., Ltd (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS101-BTC-II-1
Record Dates: First submitted 2026-01-27; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Biliary Tract Cancers (BTC)
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Injections; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cosiporfin Sodium for injection Combination Therapy Group (Experimental): Cosiporfin Sodium for injection Photodynamic Therapy Combined with Gemcitabine and Cisplatin Chemotherapy
  Interventions: Drug: Cosiporfin Sodium for injection, DVDMS; Drug: Gemcitabine Hydrochloride for Injection; Drug: Cisplatin for injection

INTERVENTIONS:
Drug: Cosiporfin Sodium for injection, DVDMS — Dosage: 0.2 mg/kg Storage: 2-8°C. Protect from light. Specifications: 10mg per bottle
Drug: Gemcitabine Hydrochloride for Injection — Specifications: 1.0g/vial, 5 vials/box Storage: Store at room temperature (15-30°C) Dosage: 1000mg/m²
Drug: Cisplatin for injection — Specifications: 20mg/vial, 8 vials/box Storage: Store in a light-protected, tightly closed container (10-30°C) Dosage: 25mg/m²

SUMMARY:
Study Design: Multicenter, open-label, Single Group Study Population: Patients with locally advanced or recurrent metastatic extrahepatic cholangiocarcinoma who are inoperable or unwilling to undergo surgery.

Primary Research Objective: To preliminarily evaluate the efficacy of photodynamic therapy (PDT) with sodium protoporphyrin combined with gemcitabine and cisplatin (GC regimen) chemotherapy in patients with advanced extrahepatic cholangiocarcinoma complicated by biliary obstruction.

Secondary Study Objective: To preliminarily evaluate the safety and tolerability of photodynamic therapy (PDT) with heme porphyrin sodium combined with gemcitabine and cisplatin (GC regimen) chemotherapy in patients with advanced extrahepatic cholangiocarcinoma with biliary obstruction.

Primary endpoint: 6-month overall survival rate (6m-OS rate)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be enrolled in this study:

  1. All subjects or their legal representatives must voluntarily sign an ethics committee-approved informed consent form in writing prior to initiating any screening procedures;
  2. Age ≥ 18 years, no gender restrictions;
  3. Patients with histologically or cytologically confirmed, locally advanced or recurrent metastatic extrahepatic cholangiocarcinoma who are inoperable or unwilling to undergo surgery;
  4. No prior systemic therapy during the recurrent or metastatic stage;
  5. Presence of obstructive lesions in the extrahepatic bile ducts, with at least one measurable lesion outside the bile ducts according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
  6. Subjects with an ECOG performance status score of 0 or 1 (see Appendix 3 for details);
  7. Subjects with an expected survival of ≥3 months;
  8. Subjects with adequate organ and bone marrow function meeting the following laboratory criteria:

     * Bone marrow function: Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L (1500/mm³) ; platelets ≥100 × 10⁹/L (1 × 10⁵/mm³); hemoglobin ≥9.0 g/dL (no treatment for bone marrow suppression, such as GCS-F, EPO, or blood transfusion, within 14 days prior to screening laboratory tests);
     * Renal Function: Creatinine clearance (Ccr) ≥50 mL/min (calculated using the Cockcroft-Gault formula; see Appendix 4);
     * Coagulation Function: International Normalized Ratio (INR) ≤1.5 × ULN; Activated Partial Thromboplastin Time (APTT) ≤1.5 × ULN;
     * Echocardiogram: Left ventricular ejection fraction (LVEF) ≥50%;
     * 12-lead electrocardiogram: Fridericia-corrected QT interval (QTcF) <470 msec (Appendix 4);
  9. Recovered from all prior treatments with toxicities resolved to Grade 1 or below;
  10. Female subjects of childbearing potential and all male subjects must agree to use highly effective contraception during the trial and for 6 months after the last dose of sodium porphyrin. contraceptive gel, contraceptive film, intrauterine device, oral or injectable contraceptives, subcutaneous implant, etc.), and women of childbearing potential must have a negative pregnancy test result within ≤7 days prior to study drug administration.

Exclusion Criteria:

* Subjects meeting any of the following criteria are ineligible for enrollment:

  1. Patients with ampullary cancer;
  2. Known hypersensitivity to sodium porphyrin or other photosensitizing agents;
  3. Diffuse liver metastases or liver tumor burden exceeding 50% of liver volume;
  4. Known or suspected brain metastases, leptomeningeal metastases, or spinal cord compression (including asymptomatic cases and those adequately treated);
  5. Subjects who participated in any other drug clinical trial or other interventional clinical trial within 4 weeks prior to study drug administration, except for subjects participating in observational (non-interventional) clinical studies or those already in the follow-up period of an interventional study;
  6. Previous exposure to photosensitizers or photodynamic therapy;
  7. Patients with unremovable stents in the extrahepatic bile ducts;
  8. Patients with prior history of immunotherapy (including but not limited to various anti-PD-1 monoclonal antibodies, anti-PD-L1 monoclonal antibodies, anti-CTLA-4 monoclonal antibodies, etc.), gemcitabine, or cisplatin treatment;
  9. Subjects who underwent major surgery within 4 weeks prior to study drug administration;
  10. Subjects who used Chinese herbal medicines with immunomodulatory or antitumor effects within 14 days prior to study drug administration;
  11. Subjects with advanced cholangiocarcinoma in a cachectic state or who are not expected to tolerate photodynamic therapy;
  12. Patients with Bismuth Type IV hilar cholangiocarcinoma;
  13. Individuals unsuitable for ERCP or endoscopic procedures;
  14. Subjects requiring concomitant antitumor therapy during study drug treatment, including chemotherapy regimens other than GC, radiotherapy, immunotherapy, or biologic agents;
  15. Any other malignancy diagnosed within 5 years prior to the first study drug administration, except for any type of carcinoma in situ, micro- or low-risk papillary thyroid carcinoma, and cured basal cell carcinoma or squamous cell carcinoma of the skin;
  16. History of allogeneic organ transplantation, or known history of autologous or allogeneic hematopoietic stem cell transplantation;
  17. Presence of clinically significant (malignant/cancerous, or moderate to large volume) pleural effusion, ascites, or pericardial effusion within 4 weeks prior to the first dose of porphyrin sodium; however, subjects with only small amounts of effusion (untreated) identified by imaging may be eligible;
  18. Presence of acute inflammation (especially necrotizing inflammation) or clinically significant active infection;
  19. Hepatitis C virus (HCV) RNA positive, active syphilis, or positive results for any one or more of the following: human immunodeficiency virus (HIV) antibody test, or active hepatitis B (defined as HBV DNA ≥ 2000 IU/mL or HBV DNA ≥ 10⁴ copies);
  20. Clinically significant cardiovascular disease or conditions, including but not limited to:

      1. Myocardial infarction within 6 months prior to first dosing;
      2. Uncontrolled angina pectoris within 3 months prior to first dosing;
      3. History or current presence of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes) or other ≥ Grade 2 persistent arrhythmias (per NCI-CTCAE v5.0);
      4. History or current presence of congestive heart failure [New York Heart Association (NYHA) Class III or IV (Appendix 5)];
      5. Complete left bundle branch block or complete right bundle branch block with left anterior fascicular block (double bundle branch block);
      6. Long QT syndrome or confirmed family history of long QT syndrome; known concomitant use of QT-prolonging medications;
      7. Bradycardia, defined as a screening ECG showing a heart rate < 45 beats per minute;
      8. Hypotension, defined as a screening systolic blood pressure ≤86 millimeters of mercury (mmHg);
      9. Uncontrolled hypertension, where the subject receives standard antihypertensive therapy but has a screening systolic blood pressure > 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg;
  21. Cerebrovascular events (including hemorrhagic, ischemic, transient ischemic attacks), cranial surgery, or unexplained loss of consciousness within 6 months prior to the first dose;
  22. Severe pre-existing conditions such as interstitial lung disease, severe dyspnea occurring at rest or requiring supplemental oxygen, inability to lie flat due to acute asthma exacerbation or respiratory failure, active or chronic liver disease, severe hepatic impairment [Child-Pugh Class C], hemorrhagic disorders secondary to hepatic insufficiency, hepatic encephalopathy, etc.; epilepsy or conditions likely to induce seizures; diseases requiring systemic immunosuppressive therapy [including immunosuppressants such as anti-TNF monoclonal antibodies, glucocorticoids (nasal inhalation or topical application permitted)]; history of adrenal insufficiency;
  23. Thromboembolic disease within 6 months prior to first dose;
  24. Uncontrolled psychiatric illness/social circumstances expected to limit compliance with study requirements or impair the subject's ability to provide written informed consent;
  25. Known history of psychiatric drug abuse or substance abuse;
  26. Pregnant or lactating women;
  27. Receipt of a live vaccine within 4 weeks prior to the first dose;
  28. Other reasons deemed by the investigator to make the subject unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
6-month overall survival rate (6m-OS rate) | Month 6

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Month 12&Month 24
Disease Control Rate (DCR) | Month 12&Month 24
Progression-Free Survival (PFS) | Month 12&Month 24
Duration of Response (DoR) | Month 12&Month 24
Overall Survival (OS) | Month 12&Month 24
12/24-Month Survival Rate | Month 12&Month 24
Time to First Chemotherapy | Month 12&Month 24
Time to Jaundice Recurrence/Recurrence Rate | Month 12&Month 24

CONTACTS AND LOCATIONS:
Locations (1):
- No. 266, Trumpet Vine Road, Shanghai, Pudong New Area, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code